CLINICAL TRIAL: NCT01398579
Title: Prospective Comparison Between Probe-based Confocal Laser Endomicroscopy, White-light Endoscopy and Virtual Chromoendoscopy for the Diagnosis of Gastric Pre-neoplastic and Neoplastic Lesions (pCLE-GCEP)
Brief Title: Comparison Between Probe-based Confocal Laser Endomicroscopy, White-light Endoscopy and Virtual Chromoendoscopy
Acronym: pCLE-GCEP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E\10\703
Record Dates: First submitted 2011-06-26; First posted 2011-07-20 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2011-08

CONDITIONS: Intestinal Metaplasia; Intestinal Dysplasia
Keywords: intestinal metaplasia; dysplasia; probe-based confocal endomicroscopy
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A: WLE followed by AFI followed by NBI followed by pCLE.
  Interventions: Procedure: Gastroscopy
- Group B (Active Comparator): Group B: WLE followed by NBI followed by AFI followed by pCLE.
  Interventions: Procedure: Gastroscopy

INTERVENTIONS:
Procedure: Gastroscopy — 20 patients will be randomized into two groups. All of them will be examined using four different endoscopy imaging technologies by one trained specialist. 10 patients will be in group A and another 10 patients will be in group B.
  Group A: WLE followed by AFI followed by NBI followed by pCLE. Group B: WLE followed by NBI followed by AFI followed by pCLE.
  Other Names: OGD

SUMMARY:
The investigators hypothesis that

1. clinical applicability and overall diagnostic sensitivity and specificity of pCLE for diagnosing gastric preneoplastic and neoplastic lesions is acceptable
2. pCLE, as compared to white-light endoscopy (WLE), AFI and magnifying NBI has higher sensitivity and specificity for the diagnosing gastric pre-neoplastic and neoplastic lesions

DETAILED DESCRIPTION:
Patients will be recruited from an ongoing study - Gastric Cancer Epidemiology, Clinical and Genetic Programme Cohort Study (GCEP). GCEP is a prospective cohort study aiming to enroll 3,000 Singapore- Chinese subjects aged >50 years, and offers screening by endoscopy and systematic follow-up for a minimum of 5 years. 20 patients will be randomized into two groups. All of them will be examined using four different endoscopy imaging technologies by one trained specialist. 10 patients will be in group A and another 10 patients will be in group B. Group A: WLE followed by AFI followed by NBI followed by pCLE. Group B: WLE followed by NBI followed by AFI followed by pCLE. The difference between two groups is the sequence of two endoscopy imaging modes - AFI and NBI. Diagnosis made during NBI and AFI must be made based on pre-defined criteria, and should not be influenced by the preceding imaging modality. To control for the possible bias on the third imaging modality caused by influence from the preceding imaging modality, patients are randomized to receive NBI before AFI or AFI before NBI.

Endoscopic diagnosis will be made for each suspected lesion with every imaging modality. The biopsy of lesions will be taken after pCLE examination is completed and sent for histology. In the absence of suspicious lesions, the area of examination will be as follows (as stated in main GCEP protocol):

* A1- lesser curvature of the antrum, within 2-3cm of the pylorus.
* A2- greater curvature of the antrum, within 2-3cm of the pylorus.
* IA- incisura angularis.
* B1- lesser curvature of the corpus, 4cm proximal to the angulus.
* B2- middle portion of the greater curvature of the corpus, 8cm from the cardia.
* Cardia (C) - within 1 cm below the OGJ (defined as the point where gastric folds disappear).

The results will be compared with the gold standard diagnosis - histopathology diagnosis. The sensitivity and specificity for each imaging tool will be calculated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* The subject is Chinese
* The subject is greater than 50 years of age
* The subject satisfies one or more of the following criteria:

  * has (had) a history of dyspepsia of at least 4 weeks or more. Dyspeptic symptoms include bloating, epigastric discomfort and early satiety
  * has a family history of gastric cancer
  * has a medical condition for which an OGD is indicated.
* Has past history of intestinal metaplasia or dysplasia
* The subject must have personally signed and dated the patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.
* The subject must be willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

* patients who cannot undergo gastroscopies
* have a personal history of stomach cancer or surgery
* any disabling illnesses
* are pregnant or breast-feeding
* have bronchial asthma or a known allergy to fluorescein
* have renal impairment with serum creatinine above the upper limit of normal
* have uncorrected coagulopathy or severe thrombocytopenia precluding biopsy
* unable to provide informed consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of accurate endoscopic diagnosis made with pCLE compared with histopathology diagnosis | An average of 1 week for which histology report will be out for comparison
  For each patient, the minimum sites of pCLE examination must consist of 2 sites at antrum, 1 site at the incisura, 2 sites at the corpus, and 1 site at the cardia. When suspicious lesions are present, more sites of pCLE examination will be allowed. Each site of pCLE examination will be biopsied and sent for histology.The pCLE examination will be video recorded and interpretation will be done independently on a separate day from the endoscopy day.The analysis will be by per biopsy site matched with corresponding video sequence

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, Prof, Principal Investigator — NUHS
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Uedo N, Ishihara R, Iishi H, Yamamoto S, Yamamoto S, Yamada T, Imanaka K, Takeuchi Y, Higashino K, Ishiguro S, Tatsuta M. A new method of diagnosing gastric intestinal metaplasia: narrow-band imaging with magnifying endoscopy. Endoscopy. 2006 Aug;38(8):819-24. doi: 10.1055/s-2006-944632. PMID 17001572
- [Background] Eisen GM, Baron TH, Dominitz JA, Faigel DO, Goldstein JL, Johanson JF, Mallery JS, Raddawi HM, Vargo JJ 2nd, Waring JP, Fanelli RD, Wheeler-Harbough J; American Society for Gastrointestinal Endoscopy. Complications of upper GI endoscopy. Gastrointest Endosc. 2002 Jun;55(7):784-93. doi: 10.1016/s0016-5107(02)70404-5. PMID 12024128
- [Result] Pohl H, Rosch T, Vieth M, Koch M, Becker V, Anders M, Khalifa AC, Meining A. Miniprobe confocal laser microscopy for the detection of invisible neoplasia in patients with Barrett's oesophagus. Gut. 2008 Dec;57(12):1648-53. doi: 10.1136/gut.2008.157461. Epub 2008 Aug 28. PMID 18755886
- [Result] Buchner AM, Shahid MW, Heckman MG, Krishna M, Ghabril M, Hasan M, Crook JE, Gomez V, Raimondo M, Woodward T, Wolfsen HC, Wallace MB. Comparison of probe-based confocal laser endomicroscopy with virtual chromoendoscopy for classification of colon polyps. Gastroenterology. 2010 Mar;138(3):834-42. doi: 10.1053/j.gastro.2009.10.053. Epub 2009 Nov 10. PMID 19909747
- [Result] Inoue T, Uedo N, Ishihara R, Kawaguchi T, Kawada N, Chatani R, Kizu T, Tamai C, Takeuchi Y, Higashino K, Iishi H, Tatsuta M, Tomita Y, Toth E. Autofluorescence imaging videoendoscopy in the diagnosis of chronic atrophic fundal gastritis. J Gastroenterol. 2010;45(1):45-51. doi: 10.1007/s00535-009-0150-7. Epub 2009 Oct 30. PMID 19876586
- [Result] Kato M, Kaise M, Yonezawa J, Yoshida Y, Tajiri H. Autofluorescence endoscopy versus conventional white light endoscopy for the detection of superficial gastric neoplasia: a prospective comparative study. Endoscopy. 2007 Nov;39(11):937-41. doi: 10.1055/s-2007-966857. PMID 18008201
- [Result] Ezoe Y, Muto M, Horimatsu T, Minashi K, Yano T, Sano Y, Chiba T, Ohtsu A. Magnifying narrow-band imaging versus magnifying white-light imaging for the differential diagnosis of gastric small depressive lesions: a prospective study. Gastrointest Endosc. 2010 Mar;71(3):477-84. doi: 10.1016/j.gie.2009.10.036. PMID 20189506
- [Result] Yao K, Iwashita A, Tanabe H, Nishimata N, Nagahama T, Maki S, Takaki Y, Hirai F, Hisabe T, Nishimura T, Matsui T. White opaque substance within superficial elevated gastric neoplasia as visualized by magnification endoscopy with narrow-band imaging: a new optical sign for differentiating between adenoma and carcinoma. Gastrointest Endosc. 2008 Sep;68(3):574-80. doi: 10.1016/j.gie.2008.04.011. Epub 2008 Jul 26. PMID 18656862
- [Result] Kato M, Kaise M, Yonezawa J, Goda K, Toyoizumi H, Yoshimura N, Yoshida Y, Kawamura M, Tajiri H. Trimodal imaging endoscopy may improve diagnostic accuracy of early gastric neoplasia: a feasibility study. Gastrointest Endosc. 2009 Nov;70(5):899-906. doi: 10.1016/j.gie.2009.03.1171. PMID 19595318
- [Result] Wallace MB, Meining A, Canto MI, Fockens P, Miehlke S, Roesch T, Lightdale CJ, Pohl H, Carr-Locke D, Lohr M, Coron E, Filoche B, Giovannini M, Moreau J, Schmidt C, Kiesslich R. The safety of intravenous fluorescein for confocal laser endomicroscopy in the gastrointestinal tract. Aliment Pharmacol Ther. 2010 Mar;31(5):548-52. doi: 10.1111/j.1365-2036.2009.04207.x. Epub 2009 Nov 30. PMID 20002025
- [Derived] Lim LG, Yeoh KG, Srivastava S, Chan YH, Teh M, Ho KY. Comparison of probe-based confocal endomicroscopy with virtual chromoendoscopy and white-light endoscopy for diagnosis of gastric intestinal metaplasia. Surg Endosc. 2013 Dec;27(12):4649-55. doi: 10.1007/s00464-013-3098-x. Epub 2013 Jul 27. PMID 23892761